CLINICAL TRIAL: NCT05063682
Title: A Phase 1 Study to Evaluate EGFRvIII -Targeted Chimeric Antigen Receptor (CAR) T Cells for Adult Patients With Leptomeningeal Glioblastoma
Brief Title: The Efficacy and Safety of Brain-targeting Immune Cells (EGFRvIII-CAR T Cells) in Treating Patients With Leptomeningeal Disease From Glioblastoma. Administering Patients EGFRvIII -CAR T Cells May Help to Recognize and Destroy Brain Tumor Cells in Patients
Acronym: CARTREMENDOUS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chembrain LTD (Industry)
Collaborators: University of Oulu (Other); Jyväskylä Central Hospital (Other); Apollo Hospital, New Delhi, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6678EGFRvIII
Record Dates: First submitted 2021-06-10; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioma, Malignant
Keywords: Glioblastoma; CAR-T; EGFRvIII
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients receive EGFRvIII -CAR T cells intracerebroventricular over 15 minutes on day 1. Patients may receive additional cycles based on the persistence of the cells.
  Interventions: Biological: EGFRvIII-specific hinge-optimized CD3 ζ-stimulatory/41BB-co-stimulatory Chimeric Antigen Receptor autologous T-lymphocytes

INTERVENTIONS:
Biological: EGFRvIII-specific hinge-optimized CD3 ζ-stimulatory/41BB-co-stimulatory Chimeric Antigen Receptor autologous T-lymphocytes — ICV administration

SUMMARY:
This phase I trial investigates the efficacy and safety of brain-targeting epidermal growth factor receptor chimeric antigen receptor immune cells (EGFRvIII-CAR T cells) in treating patients with leptomeningeal disease from glioblastoma. T cells are part of the immune system and help the body fight malignant tumours. Immune cells can be genetically modified to destroy brain tumor cells in the laboratory. EGFRvIII -CAR T cells are brain tumor specific and can enter and express its genes in immune cells. Administering patients EGFRvIII -CAR T cells may help to recognize and destroy brain tumor cells in patients with leptomeningeal disease from glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. Examine and describe the safety and feasibility of EGFRvIII-specific hinge-optimized CD3 ζ-stimulatory/41BB-co-stimulatory Chimeric Antigen Receptor autologous T-lymphocytes (EGFRvIII -CAR T cells) through intracerebroventricular (ICV) delivery as adjuvant therapy in participants with EGFRvIII+ leptomeningeal disease from glioblastoma.
2. Determine the activity of EGFRvIII -CAR T cells based on survival rate at 12 months for both arms.

SECONDARY OBJECTIVES:

1. Describe persistence, expansion and phenotype of endogenous and EGFRvIII -CAR T cells in peripheral blood (PB), tumor cyst fluid (TCF) and cerebral spinal fluid (CSF) at applicable time points
2. Describe cytokine levels in PB, TCF, and CSF at applicable time points
3. Estimate the rate of disease response by Response Assessment in Neuro-Oncology Leptomeningeal Metastases (RANO LM) criteria
4. Estimate rate of progression free survival at 6 months. Estimate rate of overall survival (OS) at 12 months by study arm.
5. Estimate time to next treatment
6. Evaluate EGFRvIII -CAR T cell persistence in the tumor tissue and the location of the EGFRvIII -CAR T cells with respect to the infusion site.
7. Evaluate biomarkers and cytokine levels

OUTLINE:

Patients receive EGFRvIII -CAR T cells intracerebroventricular over 15 minutes on day 1. Patients may receive additional cycles based on the persistence of the cells. The patients are followed extensively according to the clinical pharmacology sampling plan; on days 1-30, months 2-12, and three times per year up to 10 years based on response

ELIGIBILITY:
Inclusion Criteria:

* Participant has been treated for leptomeningeal metastases after intrathecal chemotherapy and/or radiation OR refuses to undergo additional radiation and/or intrathecal chemotherapy
* Participant must have a Karnofsky performance status (KPS) >= 60
* Participant must have a life expectancy of >= 2 months
* Women of child-bearing potential must have negative serum pregnancy test and agree to use a reliable form of birth control prior to study entry and for at least two months following study treatment. Male research participants must agree to use a reliable form of birth control and not donate sperm during the study and for at least two months following study treatment
* Participant has a histologically confirmed EGFRvII+ (epidermal growth factor receptor) tumor expression by immunohistochemistry (IHC) at the initial tumor presentation or recurrent disease (H-score >= 50)
* Participant or legal guardian must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Research participant requires supplemental oxygen to keep saturation greater than 95%
* Research participant requires dialysis
* Research participant has uncontrolled seizure activity and/or clinically evident progressive encephalopathy
* Failure of research participant or legal guardian to understand the basic elements of the protocol and/or the risks/benefits of participating in the study.
* Participant is unwilling to stop treatment with chemotherapy or endocrine therapy and/or radiation one week prior and during the first 4 cycles of the study
* Participant has ventriculoperitoneal shunt
* Participant has a coagulopathy or bleeding disorder
* Participant is HIV+ (human immunodeficiency virus) or has acute CMV (cytomegalovirus) infection
* Participant has any uncontrolled illness, including ongoing or active infection; participant has known active hepatitis B or C infection; participants with any signs or symptoms of active infection, positive blood cultures or radiological evidence of infections
* Participant has an autoimmune disease that requires constant treatment
* Participant has another active malignancy
* Participant is unable to undergo a brain magnetic resonance imaging (MRI)
* Participant is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 10 years
  Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Overall survival | 12 months

SECONDARY OUTCOMES:
CAR (chimeric antigen receptor) T cell levels detected in tumor cyst fluid (TCF), peripheral blood (PB), and cerebrospinal fluid (CSF) | Up to 6 cycles (3 months), at the end of each cycle 1 (each cycle is 14 days)
  Measured by absolute number per ul by flow
Endogenous T cell levels detected in tumor cyst fluid (TCF), peripheral blood (PB), and cerebrospinal fluid (CSF) | Up to 6 cycles (3 months), at the end of each cycle 1 (each cycle is 14 days)
  Measured by absolute number per ul by flow
Cell phenotype detected in tumor cyst fluid (TCF), peripheral blood (PB), and cerebrospinal fluid (CSF) | Up to 6 cycles (3 months), at the end of each cycle 1 (each cycle is 14 days)
  Measured by absolute number per ul by flow
Cytokine levels (Procartaplex panel) in PB, TCF and CSF | Up to 6 cycles (3 months), at the end of each cycle 1 (each cycle is 14 days)
Disease response | Up to 10 years
  Measured by Response Assessment in Neuro-Oncology Criteria (RANO LM).
Time to progression | Up to 10 years
  Progression defined by RANO LM criteria
Overall survival | Up to 10 years
CAR T and endogenous cells detected in tumor tissue | Baseline and additional time points according to response (through study completion, up to 10 years by as needed basis)
  Detected in tumor tissue by immunohistochemistry (IHC)
EGFRvII (epidermal growth factor receptor) antigen expression levels in tumor tissue. | Baseline and additional time points according to response (through study completion, up to 10 years by as needed basis)
  Descriptive statistics will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Kai Reinikainen, MD/PhD, Principal Investigator — Chembrain LTD
Locations (3):
- Finland (2):
  - Jyväskylä Central Hospital, Jyväskylä
  - University Of Oulu, Oulu
- Apollo Hospital, New Delhi, India

IPD SHARING:
Plan to Share IPD: No